CLINICAL TRIAL: NCT03851705
Title: A Two-Part (Double-Blind Placebo Controlled/Open-Label) Multicenter Study to Evaluate Safety, Tolerability, and Efficacy of Inclisiran in Subjects With Homozygous Familial Hypercholesterolemia (Hofh) (ORION-5)
Brief Title: A Study of Inclisiran in Participants With Homozygous Familial Hypercholesterolemia (HoFH)
Acronym: ORION-5
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDCO-PCS-17-02; CKJX839A12302 (Other: Novartis Pharmaceuticals); 2018-000893-31 (EudraCT Number)
Record Dates: First submitted 2019-02-07; First posted 2019-02-22 (Actual); Results first posted 2022-11-10 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Homozygous Familial Hypercholesterolemia
Keywords: HoFH
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — Injections; ALN-PCS

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 - Inclisiran (Experimental): Participants who received a dose of 300 milligram (mg) inclisiran sodium for injection administered by SC injection on Day 1 and Day 90.
  Interventions: Drug: Inclisiran Sodium for injection
- Part 1 - Placebo (Placebo Comparator): Participants who received a dose of placebos administered by SC injection on Day 1 and Day 90.
  Interventions: Drug: Placebo; Drug: Placebos
- Part 2 - Inclisiran (Experimental): Participants who received a dose of 300 mg inclisiran sodium for injection administered by SC injection on Day 270, Day 450 and Day 630. In addition, participants who were assigned to the placebo arm in Part 1 will receive a dose of 300 mg inclisiran sodium administered by SC injection on Day 180 after completion of Part 1.
  Interventions: Drug: Inclisiran Sodium for injection

INTERVENTIONS:
Drug: Inclisiran Sodium for injection — Inclisiran is a synthetic, chemically modified small interfering ribonucleic acid (siRNA) targeting proprotein convertase subtilisin kexin type 9 (PCSK9) messenger ribonucleic acid (mRNA) with a covalently attached triantennary N-acetylgalactosamine (GalNAc) ligand.
  Other Names: ALN-PCSSC; KJX839; ALN-PCSSC
  Arms: Part 1 - Inclisiran; Part 2 - Inclisiran
Drug: Placebo — Sterile normal saline (0.9% sodium chloride in water for injection)
  Arms: Part 1 - Placebo
Drug: Placebos — Sterile normal saline (0.9% sodium chloride in water for injection)
  Arms: Part 1 - Placebo

SUMMARY:
This study was a Phase III,A two-part (double-blind placebo-controlled/open-label) multicenter study to evaluate safety, tolerability, and efficacy of inclisiran in subjects with homozygous familial hypercholesterolemia (HoFH).

DETAILED DESCRIPTION:
This study had two sequential parts:

* Part 1: 6-month double-blind period in which subjects were randomized to receive either inclisiran or placebo
* Part 2: 18-month open-label follow-up period; placebo-treated subjects from Part 1 were transitioned to inclisiran at Day 180 and all subjects who participated in an open-label follow-up period of inclisiran only

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HoFH by genetic confirmation or a clinical diagnosis based on a history of an untreated LDL-C concentration >500 mg/dL (13 mmol/L) together with either xanthoma before 10 years of age or evidence of heterozygous familial hypercholesterolemia in both parents
2. Stable on a low-fat diet.
3. Subjects on statins should be receiving a maximally tolerated dose. Maximum tolerated dose is defined as the maximum dose of statin that can be taken on a regular basis without intolerable adverse events.
4. Subjects not receiving statins must have documented evidence of intolerance to at least two different statins.
5. Subjects on lipid-lower therapies (such as statin and/or ezetimibe) should be on a stable dose for ≥30 days before screening with no planned medication or dose change during study participation.
6. Fasting central laboratory LDL-C concentration ≥130 mg/dL (3.4 mmol/L).
7. Triglyceride concentration <400 mg/dL (4.5 mmol/L)
8. No current or planned renal dialysis or renal transplantation
9. Subjects on a documented regimen of LDL or plasma apheresis will be allowed to continue the apheresis during the study, if needed.
10. Subjects must be willing and able to give written informed consent before initiation of any study-related procedures. The subject should be willing to comply with all required study procedures.
11. Willing to follow all study procedures including adherence to dietary guidelines, study visits, fasting blood draws, and compliance with study treatment regimens.

Exclusion Criteria:

1. Use of Mipomersen or Lomitapide therapy within 5 months of screening
2. Treatment (within 90 days of screening) with monoclonal antibodies directed towards PCSK9
3. New York Heart Association (NYHA) class IV heart failure or last known left ventricular ejection fraction <25%
4. Major adverse cardiovascular event within 3 months prior to randomization
5. Planned cardiac surgery or revascularization
6. Uncontrolled severe hypertension: systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg prior to randomization despite anti-hypertensive therapy
7. Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or unexplained alanine aminotransferase (ALT), aspartate aminotransferase (AST), elevation >3x ULN, or total bilirubin >2x upper limit of normal (ULN) at screening confirmed by a repeat measurement at least 1 week apart
8. Severe concomitant noncardiovascular disease that carries the risk of reducing life expectancy to less than the duration of the trial
9. History of malignancy that required surgery (excluding local and wide-local excision), radiation therapy and/or commencement of systemic therapy as treatment during the 3 years prior to randomization
10. Females who are pregnant or nursing, or who are of childbearing potential and unwilling to use at least one acceptable effective method of contraception (eg, oral contraceptives, barrier methods, approved contraceptive implant, long- term injectable contraception, intrauterine device) for the entire duration of the study. Exemptions from this criterion:

    1. Women >2 years postmenopausal (defined as 1 year or longer since their last menstrual period) AND more than 55 years of age
    2. Postmenopausal women (as defined above) and less than 55 years of age with a negative pregnancy test within 24 hours of enrolment
    3. Women who are surgically sterilized at least 3 months prior to enrolment
11. Known history of alcohol and/or drug abuse within 5 years
12. Any condition that according to the investigator could interfere with the conduct of the study, such as but not limited to:

    1. Subjects who are unable to communicate or to cooperate with the investigator.
    2. Unable to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study (including subjects whose cooperation is doubtful due to drug abuse or alcohol dependency)
    3. Unlikely to comply with the protocol requirements, instructions, and study-related restrictions (eg, uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study)
    4. Have any medical or surgical condition, which in the opinion of the investigator would put the subject at increased risk from participating in the study
    5. Persons directly involved in the conduct of the study
13. Any uncontrolled or serious disease, or any medical or surgical condition, that may either interfere with participation in the clinical study, and/or put the subject at significant risk (according to investigator's [or delegate] judgment) if he/she participates in the clinical study
14. Any underlying known disease, or surgical, physical, or medical condition that, in the opinion of the Investigator, might interfere with the interpretation of clinical study results
15. Treatment with other investigational medicinal products or devices within 30 days or 5 half-lives of the screening visit, whichever is longer
16. Previous participation in the study
17. Hypersensitivity to any of the ingredients of Inclisiran

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- (50852-001) Queen Mary Hospital, Hong Kong, Hong Kong
- (50972-001) Hadassah Hospital Lipid Research Ein Kerem, Jerusalem, Israel
- Russia (3):
  - (50007-001) Research Institute of Complex Issues of Cardiovascular Diseases, Kemerovo
  - (50007-003) National Medical Research Centre of Cardiology, Moscow
  - (50007-002) Hospital for War Veterans, Saint Petersburg
- (50381-001) Clinical Center of Serbia, Belgrade, Serbia
- (50027-001) Johannesburg Hospital, Johannesburg, South Africa
- (50886-001) Taipei Veterans General Hospital, Taipei, Taiwan
- Turkey (Türkiye) (3):
  - (50090-002) University of Health Sciences, Etlik
  - (50090-003) Istanbul University, Istanbul
  - (50090-001) Ege Universitesi, Izmir
- Ukraine (2):
  - (50380-002) IMunicipal Non-commercial Enterprise "Ivano-Frankivsk Regional Clinical Cardiology Center Ivano-Frankivsk Regional Council", Ivano-Frankivsk
  - (50380-001) National Scientific Center, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- [Derived] Raal F, Durst R, Bi R, Talloczy Z, Maheux P, Lesogor A, Kastelein JJP; ORION-5 Study Investigators. Efficacy, Safety, and Tolerability of Inclisiran in Patients With Homozygous Familial Hypercholesterolemia: Results From the ORION-5 Randomized Clinical Trial. Circulation. 2024 Jan 30;149(5):354-362. doi: 10.1161/CIRCULATIONAHA.122.063460. Epub 2023 Oct 18. PMID 37850379
- [Derived] Warden BA, Duell PB. Inclisiran: A Novel Agent for Lowering Apolipoprotein B-containing Lipoproteins. J Cardiovasc Pharmacol. 2021 Aug 1;78(2):e157-e174. doi: 10.1097/FJC.0000000000001053. PMID 33990512
- See also: A Plain Language Trial Summary is available on novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1197

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 56 subjects were enrolled and 53 subjects completed through Day 180 (Part 1) and went into the Open-Label period (Part 2), in which 47 subjects completed.
Groups:
- Part 2 - Placebo-Inclisiran; Part 2 - Inclisiran-Inclisiran: Participants who received a dose of 300 mg inclisiran sodium for injection administered by SC injection on Day 270, Day 450 and Day 630. In addition, participants who were assigned to the placebo arm in Part 1 received a dose of 300 mg inclisiran administered by SC injection on Day 180 after completion of Part 1.
Period: Part 1: Double-Blind Period
Arm/Group | Part 1 - Inclisiran | Part 1 - Placebo | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Started | 37 | 19 | 0 | 0
Completed | 34 | 19 | 0 | 0
Not Completed | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Other reason | 1 | 0 | 0 | 0
Period: Part 2: Open-Label Period
Arm/Group | Part 1 - Inclisiran | Part 1 - Placebo | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Started | 0 | 0 | 34 | 19
Completed | 0 | 0 | 29 | 18
Not Completed | 0 | 0 | 5 | 1
Not completed — Other reason | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Inclisiran: Participants who received a dose of inclisiran sodium for injection administered by sub-cutaneous (SC) injection
- Placebo: Participants who received a dose of placebo administered by sub-cutaneous (SC) injection
- Total: Total of all reporting groups
Arm/Group | Inclisiran | Placebo | Total
Number analyzed (Participants) | 37 | 19 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 19 | 53
  >=65 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 11 | 34
  Male | 14 | 8 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 31 | 17 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 150
Description: Percentage Change in LDL-C levels from Baseline to Day 150
Time Frame: Baseline, Day 150
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Percentage change | 2.39 [-19.98 to 24.75] | 0.70 [-14.03 to 15.44]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Test type: Superiority; p = 0.9047, ANCOVA — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -1.68, 95% CI 2-sided [-29.19 to 25.83]

2. Secondary Outcome: Absolute Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Day 150
Description: Absolute Change in LDL-C levels (mg/dL) from baseline to Day 150
Time Frame: Baseline, Day 150
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
mg/dL | -8.82 [-75.19 to 57.55] | -2.35 [-36.34 to 31.63]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Test type: Superiority; p = 0.8685, ANCOVA — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 6.47, 95% CI 2-sided [-70.11 to 83.05]

3. Secondary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Subsequent Visits up to Day 180
Description: Percentage Change in LDL-C levels from baseline to subsequent visits on Days 90, 150, and 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Percentage change
  Day 90 | 3.3 [-13.0 to 19.6] | -8.7 [-20.3 to 2.8]
  Day 150 | -2.9 [-22.6 to 16.9] | 1.8 [-12.5 to 16.1]
  Day 180 | -1.5 [-17.0 to 14.1] | -7.2 [-19.0 to 4.6]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.2347, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -12.1, 95% CI 2-sided [-32.2 to 8.1]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.7058, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 4.6, 95% CI 2-sided [-19.9 to 29.2]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.5653, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-25.5 to 14.1]

4. Secondary Outcome: Percent Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Subsequent Visits up to Day 720
Description: Percentage Change in LDL-C levels from baseline to subsequent visits up to Day 720
Time Frame: Baseline, Days 270, 330, 450, 510, 630, 690, and 720
Population: ITT Population (Part 2): The overall number of participants analyzed represents the intent-to-treat (ITT) population. The number analyzed per row represents participants with data at each time point.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
Percentage change
  Day 270: number analyzed (Participants) | 15 | 28
  Day 270 | -10.1 (41.62) | -9.1 (33.99)
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | -14.4 (32.62) | -4.8 (50.45)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | -6.7 (26.69) | -4.7 (46.92)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | -9.3 (29.52) | 2.4 (61.70)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | -16.6 (20.45) | -6.6 (43.75)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | -8.7 (32.17) | -4.2 (42.39)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | -14.6 (26.11) | -6.2 (47.29)

5. Secondary Outcome: Absolute Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Subsequent Visits up to Day 180
Description: Absolute change in LDL-C levels (mg/dL) from baseline to subsequent visits on Days 90, 150 and 180 based on the
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
mg/dL
  Day 90 | 3.6 [-39.6 to 46.8] | -16.3 [-47.0 to 14.4]
  Day 150 | -17.2 [-70.8 to 36.3] | 0.5 [-38.3 to 39.2]
  Day 180 | -7.0 [-50.5 to 36.4] | -14.5 [-47.5 to 18.5]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.4589, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -19.9, 95% CI 2-sided [-73.3 to 33.6]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.5956, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 17.7, 95% CI 2-sided [-48.8 to 84.3]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.7861, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -7.5, 95% CI 2-sided [-62.7 to 47.7]

6. Secondary Outcome: Absolute Change in Low-Density Lipoprotein Cholesterol (LDL-C) From Baseline to Subsequent Visits up to Day 720
Description: Absolute change in LDL-C levels from Baseline to Subsequent Visits up to Day 720
Time Frame: Baseline, Days 270, 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
mg/dL
  Day 270: number analyzed (Participants) | 15 | 28
  Day 270 | -27.3 (154.94) | -17.5 (85.85)
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | -37.2 (123.09) | -17.9 (113.10)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | -12.3 (108.49) | -19.8 (111.41)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | -20.9 (118.05) | -2.2 (127.13)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | -50.5 (70.47) | -14.9 (107.90)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | -27.9 (115.46) | -8.6 (112.93)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | -43.5 (92.99) | -11.0 (124.27)

7. Secondary Outcome: Percent Change in Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) From Baseline to Subsequent Visits up to Day 180
Description: Percentage Change in PCSK9 from baseline to subsequent visits up to Day 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Percentage change
  Day 90 | 9.1 [-5.1 to 23.3] | -53.5 [-63.6 to -43.3]
  Day 150 | 4.1 [-14.3 to 22.6] | -56.5 [-69.9 to -43.1]
  Day 180 | 39.2 [17.0 to 61.5] | -53.1 [-70.2 to -35.9]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p < .0001, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -62.6, 95% CI 2-sided [-80.1 to -45.1]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p < .0001, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -60.6, 95% CI 2-sided [-83.5 to -37.8]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p < .0001, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -92.3, 95% CI 2-sided [-120.4 to -64.2]

8. Secondary Outcome: Percent Change in Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) From Baseline to Subsequent Visits up to Day 720
Description: Percentage Change in PCSK9 from baseline to subsequent visits up to Day 720
Time Frame: Baseline, Days 270, 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
Percentage Change
  Day 270: number analyzed (Participants) | 15 | 28
  Day 270 | -21.5 (55.71) | -14.4 (160.60)
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | -42.6 (32.08) | -57.0 (30.36)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | -35.8 (37.55) | -51.1 (27.90)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | -54.0 (23.62) | -59.4 (24.13)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | -41.7 (29.19) | -48.1 (32.65)
  Day 690: number analyzed (Participants) | 14 | 20
  Day 690 | -48.3 (22.30) | -64.3 (11.21)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | -53.8 (16.66) | -57.6 (39.76)

9. Secondary Outcome: Absolute Change in Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) From Baseline to Subsequent Visits up to Day 180
Description: Absolute Change in PCSK9 from baseline to subsequent visits up to Day 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: ug/L
Groups:
- Part 1 - Placebo: Participants will receive a dose of placebos administered by SC injection on Day 1 and Day 90.
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
ug/L
  Day 90 | -25.8 [-110.3 to 58.6] | -342.5 [-403.0 to -282.0]
  Day 150 | -30.7 [-114.4 to 52.9] | -335.2 [-396.1 to -274.3]
  Day 180 | 88.8 [-1.2 to 178.9] | -301.5 [-371.4 to -231.7]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p < .0001, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -316.6, 95% CI 2-sided [-420.7 to -212.6]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p < .0001, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -304.4, 95% CI 2-sided [-408.0 to -200.8]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p < .0001, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -390.4, 95% CI 2-sided [-504.5 to -276.3]

10. Secondary Outcome: Absolute Change in Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) From Baseline to Subsequent Visits up to Day 720
Description: Absolute Change in PCSK9 from baseline to subsequent visits up to Day 720
Time Frame: Baseline, Days 270, 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
ug/L
  Day 270: number analyzed (Participants) | 15 | 28
  Day 270 | -174.7 (252.10) | -234.4 (242.25)
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | -232.1 (193.51) | -392.0 (422.93)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | -237.5 (199.34) | -387.6 (483.81)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | -304.8 (181.41) | -381.0 (261.04)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | -243.6 (201.07) | -303.1 (200.37)
  Day 690: number analyzed (Participants) | 14 | 20
  Day 690 | -275.5 (163.85) | -441.8 (278.87)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | -296.8 (171.96) | -413.2 (460.33)

11. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Subsequent Visits up to Day 180
Description: Percentage change in total cholesterol from baseline to subsequent visits up to Day 180
Time Frame: Baseline, Days 90, 150 and 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Percentage Change
  Day 90 | 2.0 [-11.0 to 14.9] | -5.9 [-15.1 to 3.3]
  Day 150 | -1.5 [-17.2 to 14.1] | 1.2 [-10.1 to 12.5]
  Day 180 | -1.4 [-13.8 to 11.0] | -4.9 [-14.3 to 4.5]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.3299, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -7.9, 95% CI 2-sided [-23.9 to 8.2]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.7778, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 2.7, 95% CI 2-sided [-16.7 to 22.2]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.6613, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-19.2 to 12.3]

12. Secondary Outcome: Absolute Change in Total Cholesterol From Baseline to Subsequent Visits up to Day 180
Description: Absolute Change in total cholesterol from baseline to subsequent visits up to Day 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
mg/dL
  Day 90 | 3.9 [-40.6 to 48.4] | -15.1 [-46.7 to 16.4]
  Day 150 | -10.5 [-65.5 to 44.5] | 0.6 [-39.2 to 40.4]
  Day 180 | -6.8 [-51.7 to 38.1] | -12.6 [-46.6 to 21.3]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.4911, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -19.0, 95% CI 2-sided [-74.0 to 36.0]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.7461, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 11.1, 95% CI 2-sided [-57.2 to 79.4]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.8370, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -5.9, 95% CI 2-sided [-62.8 to 51.1]

13. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Subsequent Visits up to Day 720
Description: Percentage change in total cholesterol from baseline to subsequent visits up to Day 720
Time Frame: Baseline, Days 270, 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
Percentage Change
  Day 270: number analyzed (Participants) | 15 | 28
  Day 270 | -7.4 (34.80) | -4.8 (27.31)
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | -10.9 (27.67) | -1.0 (39.20)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | -4.2 (22.45) | -2.2 (36.05)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | -6.4 (25.37) | 2.8 (46.77)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | -11.9 (17.58) | -4.8 (33.84)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | -6.2 (26.71) | -1.9 (33.83)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | -11.2 (21.86) | -2.9 (36.70)

14. Secondary Outcome: Absolute Change in Total Cholesterol From Baseline to Subsequent Visits up to Day 720
Description: Absolute Change in total cholesterol from baseline to subsequent visits up to Day 720
Time Frame: Baseline, Days 270, 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
mg/dL
  Day 270: number analyzed (Participants) | 15 | 28
  Day 270 | -24.9 (154.60) | -13.3 (90.68)
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | -35.6 (127.19) | -13.0 (115.59)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | -7.9 (107.22) | -14.4 (113.71)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | -17.8 (120.40) | 0.1 (128.73)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | -44.5 (71.81) | -14.9 (111.50)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | -21.6 (118.21) | -6.9 (114.58)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | -40.4 (93.21) | -8.5 (126.48)

15. Secondary Outcome: Percent Change in Apolipoprotein B (apoB) From Baseline to Subsequent Visits up to Day 180
Description: Percentage change in Apolipoprotein B (apoB) from baseline to subsequent visits up to Day 180 demonstrated by Mixed Model Repeated Measures statisitical method.
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Percentage change
  Day 90 | 6.3 [-7.3 to 19.9] | -6.4 [-16.1 to 3.3]
  Day 150 | 2.8 [-12.5 to 18.1] | -0.7 [-11.8 to 10.3]
  Day 180 | 4.5 [-8.9 to 17.9] | -5.8 [-15.9 to 4.3]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.1371, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -12.7, 95% CI 2-sided [-29.5 to 4.2]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.7100, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-22.6 to 15.5]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.2278, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -10.3, 95% CI 2-sided [-27.2 to 6.6]

16. Secondary Outcome: Percent Change in Apolipoprotein B (apoB) From Baseline to Subsequent Visits up to Day 720
Description: Percentage Change in Apolipoprotein B (apoB) from baseline to subsequent visits up to Day 720
Time Frame: Baseline, Days 270, 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
Percentage Change
  Day 270: number analyzed (Participants) | 15 | 28
  Day 270 | -0.6 (40.91) | -3.3 (28.67)
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | -7.9 (28.56) | -3.6 (34.35)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | -1.3 (21.62) | -3.5 (35.66)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | -3.7 (24.21) | 1.9 (44.49)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | -7.3 (17.81) | -6.6 (32.97)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | -3.7 (27.16) | -5.8 (32.38)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | -10.4 (19.68) | -8.0 (31.93)

17. Secondary Outcome: Absolute Change in Apolipoprotein B (apoB) From Baseline to Subsequent Visits up to Day 180
Description: Absolute change in Apolipoprotein B (apoB) from baseline to subsequent visits up to Day 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
mg/dL
  Day 90 | 10.0 [-14.5 to 34.5] | -9.4 [-26.8 to 8.0]
  Day 150 | 3.3 [-24.9 to 31.6] | -1.4 [-21.9 to 19.0]
  Day 180 | 8.4 [-16.5 to 33.3] | -7.4 [-26.2 to 11.4]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.2044, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -19.4, 95% CI 2-sided [-49.7 to 10.9]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.7875, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -4.8, 95% CI 2-sided [-39.9 to 30.4]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.3193, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -15.8, 95% CI 2-sided [-47.3 to 15.7]

18. Secondary Outcome: Absolute Change in Apolipoprotein B (Apo B) From Baseline to Subsequent Visits up to Day 720
Description: Absolute Change in Apolipoprotein B (Apo B) from baseline to subsequent visits up to Day 720
Time Frame: Baseline, Days 270, 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
mg/dL
  Day 270: number analyzed (Participants) | 15 | 28
  Day 270 | -1.3 (83.72) | -1.9 (51.79)
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | -11.5 (66.78) | -7.3 (56.52)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | 3.0 (53.54) | -6.9 (61.89)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | -3.5 (58.45) | 1.1 (70.40)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | -15.4 (38.17) | -10.1 (57.06)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | -10.6 (61.77) | -10.3 (54.82)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | -22.1 (45.29) | -13.0 (55.14)

19. Secondary Outcome: Percent Change in Non-HDL Cholesterol (Non-HDL-C) From Baseline to Subsequent Visits up to Day 180
Description: Percentage change in non-HDL-C levels from baseline to subsequent visits up to Day 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Percentage change
  Day 90 | 2.9 [-12.4 to 18.2] | -7.2 [-18.1 to 3.6]
  Day 150 | -1.7 [-19.9 to 16.6] | 1.3 [-11.9 to 14.5]
  Day 180 | -1.1 [-15.6 to 13.3] | -6.2 [-17.1 to 4.7]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.2877, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -10.1, 95% CI 2-sided [-29.0 to 8.8]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.7944, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 3.0, 95% CI 2-sided [-19.7 to 25.7]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.5803, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-23.4 to 13.3]

20. Secondary Outcome: Percent Change in Non-HDL Cholesterol (Non-HDL-C) From Baseline to Subsequent Visits up to Day 720
Description: Percentage Change in non-HDL-C from Baseline to subsequent visits up to Day 720
Time Frame: Baseline, Days 270, 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
Percentage Change
  Day 270: number analyzed (Participants) | 15 | 28
  Day 270 | -8.4 (39.76) | -7.6 (30.95)
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | -13.1 (31.27) | -2.3 (45.56)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | -5.5 (25.49) | -3.1 (43.73)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | -8.0 (28.00) | 2.0 (55.28)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | -13.6 (18.88) | -6.5 (40.16)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | -6.4 (30.12) | -3.6 (40.11)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | -12.3 (23.99) | -5.0 (43.40)

21. Secondary Outcome: Absolute Change in Non-HDL Cholesterol (Non-HDL-C) From Baseline to Subsequent Visits up to Day 180
Description: Absolute change in non-HDL-C levels from Baseline to subsequent visits up to Day 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
mg/dL
  Day 90 | 3.8 [-40.3 to 47.8] | -15.3 [-46.5 to 15.9]
  Day 150 | -11.6 [-66.4 to 43.3] | 0.6 [-39.1 to 40.3]
  Day 180 | -5.7 [-50.2 to 38.9] | -12.7 [-46.4 to 21.0]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.4848, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -19.1, 95% CI 2-sided [-73.6 to 35.3]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.7220, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 12.2, 95% CI 2-sided [-56.0 to 80.3]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.8036, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -7.0, 95% CI 2-sided [-63.6 to 49.5]

22. Secondary Outcome: Absolute Change in Non-HDL Cholesterol (Non-HDL-C) From Baseline to Subsequent Visits up to Day 720
Description: Absolute Change in non-HDL Cholesterol (non-HDL-C) from Baseline to Subsequent Visits up to Day 720
Time Frame: Baseline, Days 270, 330, 450, 510, 630, 690, and 720
Population: ITT Population (Part 2): The overall number of participants analyzed represents the intent-to-treat (ITT) population. The number analyzed per row represents participants with data at each time point.
  .
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
mg/dL
  Day 270: number analyzed (Participants) | 15 | 28
  Day 270 | -24.7 (157.98) | -17.1 (86.34)
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | -37.2 (127.12) | -13.9 (114.51)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | -8.8 (109.91) | -15.8 (112.63)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | -19.3 (120.58) | -2.4 (128.45)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | -43.8 (70.56) | -14.7 (112.04)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | -21.0 (116.12) | -7.8 (114.44)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | -38.9 (91.89) | -9.3 (127.46)

23. Secondary Outcome: Individual Responsiveness of Subjects: Part 1
Description: Individual Responsiveness of Subjects defined as the number of subjects reaching on treatment LDL-C levels of <25 mg/dL, <50 mg/dL, <70 mg/dL, and <100 mg/dL up to Day 180
Time Frame: Days 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population. The number analyzed per row represents participants with data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Participants
  <25 mg/dL- Day 150: number analyzed (Participants) | 18 | 34
  <25 mg/dL- Day 150 | 0 | 0
  <50 mg/dL- Day 150: number analyzed (Participants) | 18 | 34
  <50 mg/dL- Day 150 | 1 | 0
  <70 mg/dL- Day 150: number analyzed (Participants) | 18 | 34
  <70 mg/dL- Day 150 | 1 | 2
  <100 mg/dL- Day 150: number analyzed (Participants) | 18 | 34
  <100 mg/dL- Day 150 | 1 | 5
  >= 100 mg/dL- Day 150: number analyzed (Participants) | 18 | 34
  >= 100 mg/dL- Day 150 | 17 | 29
  <25 mg/dL- Day 180: number analyzed (Participants) | 19 | 31
  <25 mg/dL- Day 180 | 0 | 0
  <50 mg/dL- Day 180: number analyzed (Participants) | 19 | 31
  <50 mg/dL- Day 180 | 0 | 1
  <70 mg/dL- Day 180: number analyzed (Participants) | 19 | 31
  <70 mg/dL- Day 180 | 0 | 2
  <100 mg/dL- Day 180: number analyzed (Participants) | 19 | 31
  <100 mg/dL- Day 180 | 0 | 5
  >= 100 mg/dL- Day 180: number analyzed (Participants) | 19 | 31
  >= 100 mg/dL- Day 180 | 19 | 26

24. Secondary Outcome: Individual Responsiveness of Subjects: Part 2
Description: Individual Responsiveness of Subjects defined as the number of subjects reaching on treatment LDL-C levels of <25 mg/dL, <50 mg/dL, <70 mg/dL, and <100 mg/dL up to Day 720
Time Frame: Days 330, 510, 690 and 720
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
Participants
  <25 mg/dL- Day 330: number analyzed (Participants) | 16 | 25
  <25 mg/dL- Day 330 | 0 | 0
  <50 mg/dL- Day 330: number analyzed (Participants) | 16 | 25
  <50 mg/dL- Day 330 | 1 | 0
  <70 mg/dL- Day 330: number analyzed (Participants) | 16 | 25
  <70 mg/dL- Day 330 | 2 | 1
  <100 mg/dL- Day 330: number analyzed (Participants) | 16 | 25
  <100 mg/dL- Day 330 | 2 | 5
  >= 100 mg/dL- Day 330: number analyzed (Participants) | 16 | 25
  >= 100 mg/dL- Day 330 | 14 | 20
  <25 mg/dL- Day 510: number analyzed (Participants) | 17 | 30
  <25 mg/dL- Day 510 | 0 | 0
  <50 mg/dL- Day 510: number analyzed (Participants) | 17 | 30
  <50 mg/dL- Day 510 | 0 | 2
  <70 mg/dL- Day 510: number analyzed (Participants) | 17 | 30
  <70 mg/dL- Day 510 | 0 | 3
  < 100 mg/dL- Day 510: number analyzed (Participants) | 17 | 30
  < 100 mg/dL- Day 510 | 1 | 5
  >= 100 mg/dL- Day 510: number analyzed (Participants) | 17 | 30
  >= 100 mg/dL- Day 510 | 16 | 25
  <25 mg/dL- Day 690: number analyzed (Participants) | 14 | 22
  <25 mg/dL- Day 690 | 0 | 0
  <50 mg/dL- Day 690: number analyzed (Participants) | 14 | 22
  <50 mg/dL- Day 690 | 0 | 0
  <70 mg/dL- Day 690: number analyzed (Participants) | 14 | 22
  <70 mg/dL- Day 690 | 0 | 1
  <100 mg/dL- Day 690: number analyzed (Participants) | 14 | 22
  <100 mg/dL- Day 690 | 1 | 2
  >= 100 mg/dL- Day 690: number analyzed (Participants) | 14 | 22
  >= 100 mg/dL- Day 690 | 13 | 20
  <25 mg/dL- Day 720: number analyzed (Participants) | 18 | 27
  <25 mg/dL- Day 720 | 0 | 0
  <50 mg/dL- Day 720: number analyzed (Participants) | 18 | 27
  <50 mg/dL- Day 720 | 0 | 1
  <70 mg/dL- Day 720: number analyzed (Participants) | 18 | 27
  <70 mg/dL- Day 720 | 1 | 1
  <100 mg/dL- Day 720: number analyzed (Participants) | 18 | 27
  <100 mg/dL- Day 720 | 1 | 5
  >= 100 mg/dL- Day 720: number analyzed (Participants) | 18 | 27
  >= 100 mg/dL- Day 720 | 17 | 22

25. Secondary Outcome: Proportional Responsiveness: Part 1
Description: Number of participants in each group who attain global lipid targets for their indication
Time Frame: Days 150, 180
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Participants
  Day 150: number analyzed (Participants) | 18 | 34
  Day 150 | 1 | 3
  Day 180: number analyzed (Participants) | 19 | 31
  Day 180 | 0 | 3

26. Secondary Outcome: Proportional Responsiveness of Subjects: Part 2
Description: Number of participants in each group who attain global lipid targets for their indication
Time Frame: Days 330, 510, 690 and 720
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
Participants
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | 2 | 2
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | 0 | 4
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | 0 | 1
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | 1 | 2

27. Secondary Outcome: LDL-C Reduction ≥20% or ≥30% From Baseline: Part 1
Description: Proportion of subjects in each group with ≥20% or ≥30% LDL-C reduction from Baseline in Part 1 (Days 90, 150, 180)
Time Frame: Baseline, Days 90, 150, 180
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Inclisiran | Part 1 - Placebo
Number analyzed (Participants) | 19 | 37
Participants
  LDL-C >=20%: Day 90 | 4 | 14
  LDL-C >=20%: Day 150: number analyzed (Participants) | 18 | 34
  LDL-C >=20%: Day 150 | 3 | 9
  LDL-C >=20%: Day 180: number analyzed (Participants) | 19 | 31
  LDL-C >=20%: Day 180 | 3 | 12
  LDL-C >=30%: Day 90 | 3 | 13
  LDL-C >=30%: Day 150: number analyzed (Participants) | 18 | 34
  LDL-C >=30%: Day 150 | 3 | 6
  LDL-C >=30%: Day 180: number analyzed (Participants) | 19 | 31
  LDL-C >=30%: Day 180 | 2 | 10

28. Secondary Outcome: LDL-C Reduction ≥20% or ≥30% From Baseline: Part 2
Description: Proportion of subjects in each group with ≥20% or ≥30% LDL-C reduction from Baseline in Part 2 (Days 330, 510, 690, and 720)
Time Frame: Baseline, Days 330, 510, 690, and 720
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
Participants
  LDL-C >=20%: Day 330: number analyzed (Participants) | 16 | 25
  LDL-C >=20%: Day 330 | 5 | 13
  LDL-C >=20%: Day 510: number analyzed (Participants) | 17 | 30
  LDL-C >=20%: Day 510 | 6 | 11
  LDL-C >=20%: Day 690: number analyzed (Participants) | 14 | 22
  LDL-C >=20%: Day 690 | 8 | 11
  LDL-C >=20%: Day 720: number analyzed (Participants) | 18 | 27
  LDL-C >=20%: Day 720 | 7 | 13
  LDL-C >=30%: Day 330: number analyzed (Participants) | 16 | 25
  LDL-C >=30%: Day 330 | 4 | 8
  LDL-C >=30%: Day 510: number analyzed (Participants) | 17 | 30
  LDL-C >=30%: Day 510 | 4 | 9
  LDL-C >=30%: Day 690: number analyzed (Participants) | 14 | 22
  LDL-C >=30%: Day 690 | 4 | 5
  LDL-C >=30%: Day 720: number analyzed (Participants) | 18 | 27
  LDL-C >=30%: Day 720 | 5 | 8

29. Secondary Outcome: Percent Change in High-Density Lipoprotein Cholesterol Levels (HDL-C) From Baseline to Subsequent Visits up to Day 180
Description: Percentage Change in HDL-C levels (mg/dL) from baseline to subsequent visits on Day 90, 150, and 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Percentage change
  Day 90 | -1.1 [-8.6 to 6.5] | 1.4 [-4.0 to 6.7]
  Day 150 | 2.3 [-8.0 to 12.6] | 3.6 [-3.9 to 11.1]
  Day 180 | -1.9 [-9.8 to 6.0] | 1.5 [-4.5 to 7.6]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.6028, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-6.8 to 11.7]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.8428, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-11.5 to 14.0]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.4946, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 3.4, 95% CI 2-sided [-6.6 to 13.4]

30. Secondary Outcome: Percent Change in High-Density Lipoprotein Cholesterol Levels (HDL-C) From Baseline to Subsequent Visits up to Day 720
Description: Percentage change in LDL-C levels from Baseline to Subsequent Visits up to Day 720
Time Frame: Baseline, Days 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
Percentage change
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | 3.2 (13.09) | 4.3 (16.45)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | 1.6 (12.26) | 4.8 (17.81)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | 2.9 (19.83) | 7.9 (17.75)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | -2.0 (14.81) | 0.5 (15.81)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | -2.4 (19.17) | 4.5 (20.31)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | -3.6 (14.90) | 4.1 (16.99)

31. Secondary Outcome: Absolute Change in High-Density Lipoprotein Cholesterol Levels (HDL-C) From Baseline to Subsequent Visits up to Day 180
Description: Absolute Change in HDL-C levels (mg/dL) from baseline to subsequent visits on Day 90, 150, and 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
mg/dL
  Day 90 | -0.0 [-3.4 to 3.4] | 0.2 [-2.2 to 2.6]
  Day 150 | 1.0 [-3.5 to 5.4] | -0.0 [-3.2 to 3.2]
  Day 180 | -1.2 [-4.5 to 2.1] | 0.0 [-2.5 to 2.5]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.9237, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-4.0 to 4.4]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.7177, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-6.5 to 4.5]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.5416, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-2.9 to 5.4]

32. Secondary Outcome: Absolute Change in High-Density Lipoprotein Cholesterol Levels (HDL-C) From Baseline to Subsequent Visits up to Day 720
Description: Absolute change in LDL-C levels from Baseline to Subsequent Visits up to Day 720
Time Frame: Baseline, Days 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
mg/dL
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | 1.6 (6.05) | 0.9 (6.85)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | 0.9 (6.04) | 1.4 (8.53)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | 1.5 (8.78) | 2.5 (7.86)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | -0.7 (7.35) | -0.2 (7.70)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | -0.6 (9.57) | 1.0 (8.31)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | -1.5 (7.22) | 0.8 (7.34)

33. Secondary Outcome: Absolute Change in Very-Low-Density Lipoprotein Cholesterol (VLDL-C) From Baseline to Subsequent Visits up to Day 180
Description: Absolute Change in VLDL-C levels from baseline to subsequent visits on Days 90, 150, and 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
mg/dL
  Day 90 | 0.6 [-2.8 to 4.0] | 1.6 [-0.9 to 4.0]
  Day 150 | 3.0 [-1.3 to 7.3] | 0.4 [-2.7 to 3.4]
  Day 180 | 1.8 [-3.0 to 6.5] | 1.5 [-2.1 to 5.1]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.6497, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-3.2 to 5.2]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.3209, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-7.9 to 2.6]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.9294, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-6.3 to 5.7]

34. Secondary Outcome: Absolute Change in Very-Low-Density-Lipoprotein Cholesterol Levels (VLDL-C) From Baseline to Subsequent Visits up to Day 720
Description: Absolute change in VLDL-C levels from Baseline to Subsequent Visits up to Day 720
Time Frame: Baseline, Days 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
mg/dL
  Day 330: number analyzed (Participants) | 16 | 24
  Day 330 | 0.0 (9.38) | 2.7 (8.03)
  Day 450: number analyzed (Participants) | 17 | 28
  Day 450 | 1.1 (5.84) | 4.4 (8.91)
  Day 510: number analyzed (Participants) | 16 | 30
  Day 510 | -0.9 (4.76) | -0.2 (8.85)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | 6.7 (13.76) | 0.2 (8.39)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | 6.9 (14.58) | 0.8 (9.34)
  Day 720: number analyzed (Participants) | 17 | 27
  Day 720 | 2.5 (6.81) | 1.7 (9.06)

35. Secondary Outcome: Percent Change in Very-Low-Density Lipoprotein Cholesterol (VLDL-C) From Baseline to Subsequent Visits up to Day 180
Description: Percentage Change in VLDL-C levels (mg/dL) from baseline to subsequent visits on Days 90, 150, and 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Percentage change
  Day 90 | 0.6 [-17.4 to 18.7] | 11.9 [-1.0 to 24.9]
  Day 150 | 16.3 [-1.6 to 34.1] | 4.9 [-7.8 to 17.6]
  Day 180 | 10.0 [-13.4 to 33.5] | 12.3 [-5.3 to 29.9]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.3105, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 11.3, 95% CI 2-sided [-10.8 to 33.4]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.3018, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -11.4, 95% CI 2-sided [-33.3 to 10.5]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.8755, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = 2.3, 95% CI 2-sided [-27.0 to 31.6]

36. Secondary Outcome: Percent Change in Very-Low-Density-Lipoprotein Cholesterol Levels (VLDL-C) From Baseline to Subsequent Visits up to Day 720
Description: Percentage change in VLDL-C levels from Baseline to Subsequent Visits up to Day 720
Time Frame: Baseline, Days 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
Percentage Change
  Day 330: number analyzed (Participants) | 16 | 24
  Day 330 | 6.8 (38.92) | 20.8 (57.44)
  Day 450: number analyzed (Participants) | 17 | 28
  Day 450 | 7.1 (28.86) | 23.9 (46.36)
  Day 510: number analyzed (Participants) | 16 | 30
  Day 510 | 2.1 (33.45) | 7.1 (43.16)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | 25.1 (44.22) | 6.2 (46.21)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | 26.5 (51.79) | 11.4 (59.86)
  Day 720: number analyzed (Participants) | 17 | 27
  Day 720 | 13.9 (33.26) | 12.4 (50.37)

37. Secondary Outcome: Absolute Change in Apolipoprotein A-1 (Apo-A1) mg/dL From Baseline to Subsequent Visits up to Day 180
Description: Absolute Change in Apolipoprotein A-1 (Apo-A1) from baseline to subsequent visits on Days 90, 150, and 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
mg/dL
  Day 90 | 2.6 [-5.2 to 10.3] | 0.6 [-4.9 to 6.1]
  Day 150 | 4.0 [-6.5 to 14.6] | -1.4 [-9.1 to 6.3]
  Day 180 | 1.4 [-6.9 to 9.8] | -1.3 [-7.7 to 5.1]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.6848, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-11.5 to 7.6]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.4075, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -5.4, 95% CI 2-sided [-18.5 to 7.6]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.5998, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -2.8, 95% CI 2-sided [-13.4 to 7.8]

38. Secondary Outcome: Absolute Change Apolipoprotein A-1 (Apo-A1) From Baseline to Subsequent Visits up to Day 720
Description: Absolute change in Apolipoprotein A-1 (Apo-A1) from Baseline to Subsequent Visits up to Day 720
Time Frame: Baseline, Days 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
mg/dL
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | 0.9 (14.14) | 1.2 (13.85)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | 4.9 (14.04) | 4.7 (16.59)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | 6.7 (20.39) | 7.8 (16.32)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | 5.4 (15.59) | 1.3 (13.11)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | 6.9 (17.07) | 9.3 (15.69)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | 3.9 (15.15) | 6.9 (11.30)

39. Secondary Outcome: Percent Change in Apolipoprotein A-1 (Apo-A1) From Baseline to Subsequent Visits up to Day 180
Description: Percentage Change in Apolipoprotein A-1 (Apo-A1) from baseline to subsequent visits on Day 90, 150, and 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Percentage change
  Day 90 | 1.6 [-4.5 to 7.6] | 0.6 [-3.7 to 4.9]
  Day 150 | 3.0 [-5.1 to 11.1] | 0.4 [-5.5 to 6.3]
  Day 180 | 1.6 [-5.0 to 8.3] | -1.0 [-6.1 to 4.1]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.7958, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-8.4 to 6.5]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.6003, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-12.7 to 7.4]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.5352, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -2.6, 95% CI 2-sided [-11.0 to 5.8]

40. Secondary Outcome: Percent Change Apolipoprotein A-1 (Apo-A1) From Baseline to Subsequent Visits up to Day 720
Description: Percentage change in Apolipoprotein A-1 (Apo-A1) from Baseline to Subsequent Visits up to Day 720
Time Frame: Baseline, Days 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
Percentage change
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | 0.4 (11.37) | 1.3 (10.80)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | 4.4 (10.76) | 3.9 (12.71)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | 6.2 (17.00) | 6.8 (13.40)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | 5.4 (11.11) | 0.8 (9.93)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | 5.6 (13.92) | 7.2 (12.17)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | 3.5 (11.71) | 5.5 (9.27)

41. Secondary Outcome: Percent Change in Lipoprotein(a) [Lp(a)] From Baseline to Subsequent Visits up to Day 180
Description: Percentage Change in Lp(a) from Baseline to Subsequent Visits up to Day 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Percentage change
  Day 90 | 4.3 [-6.2 to 14.7] | -4.6 [-12.2 to 2.9]
  Day 150 | 15.2 [-6.8 to 37.2] | -3.8 [-19.8 to 12.2]
  Day 180 | 4.9 [-6.5 to 16.4] | -4.8 [-13.5 to 4.0]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.1716, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -8.9, 95% CI 2-sided [-21.8 to 4.0]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.1671, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -19.0, 95% CI 2-sided [-46.2 to 8.2]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.1808, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -9.7, 95% CI 2-sided [-24.2 to 4.7]

42. Secondary Outcome: Percent Change in Lipoprotein(a) [Lp(a)] From Baseline to Subsequent Visits up to Day 720
Description: Percentage change in Lp(a) from Baseline to Subsequent Visits up to Day 720
Time Frame: Baseline, Days 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
Percentage change
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | 2.5 (33.15) | -1.4 (26.69)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | 3.4 (45.12) | 0.2 (26.42)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | 8.3 (44.74) | 13.4 (39.37)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | -8.4 (32.65) | 1.7 (29.43)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | -10.7 (34.02) | -5.3 (27.44)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | -11.4 (51.06) | -3.1 (45.08)

43. Secondary Outcome: Absolute Change in Lipoprotein(a) [Lp(a)] From Baseline to Subsequent Visits up to Day 180
Description: Absolute Change in Lp(a) from baseline to subsequent visits up to Day 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: nmol/L
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
nmol/L
  Day 90 | 5.8 [-9.4 to 20.9] | -3.8 [-14.7 to 7.1]
  Day 150 | 3.9 [-12.8 to 20.6] | -5.6 [-17.7 to 6.5]
  Day 180 | 1.2 [-12.4 to 14.7] | -5.1 [-15.3 to 5.2]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 90; Test type: Superiority; p = 0.3077, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -9.6, 95% CI 2-sided [-28.3 to 9.1]
Statistical Analysis 2: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 150; Test type: Superiority; p = 0.3628, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -9.4, 95% CI 2-sided [-30.1 to 11.2]
Statistical Analysis 3: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Day 180; Test type: Superiority; p = 0.4669, Mixed Model Repeated Measures — The a priori threshold for statistical significance was <0.05 (two-sided); Mean Difference (Final Values) = -6.2, 95% CI 2-sided [-23.2 to 10.8]

44. Secondary Outcome: Absolute Change in Lipoprotein(a) [Lp(a)] From Baseline to Subsequent Visits up to Day 720
Description: Absolute change in Lp(a) from Baseline to Subsequent Visits up to Day 720
Time Frame: Baseline, Days 330, 450, 510, 630, 690, and 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
nmol/L
  Day 330: number analyzed (Participants) | 16 | 25
  Day 330 | -3.1 (36.71) | -5.2 (30.65)
  Day 450: number analyzed (Participants) | 18 | 28
  Day 450 | -3.8 (47.48) | 3.1 (41.28)
  Day 510: number analyzed (Participants) | 17 | 30
  Day 510 | 14.5 (50.25) | 18.4 (53.31)
  Day 630: number analyzed (Participants) | 14 | 21
  Day 630 | -2.4 (31.18) | 13.7 (50.77)
  Day 690: number analyzed (Participants) | 14 | 22
  Day 690 | -5.3 (26.52) | 5.8 (26.46)
  Day 720: number analyzed (Participants) | 18 | 27
  Day 720 | -6.0 (48.12) | 5.2 (30.44)

45. Secondary Outcome: Percent Change in High-Sensitivity C-Reactive Protein (hsCRP) From Baseline to Subsequent Visits up to Day 180: Part 1
Description: Percent change in hsCRP from Baseline to subsequent visits up to Day 180
Time Frame: Baseline, Days 90, 150, 180
Population: ITT Population (Part 1): The overall number of participants analyzed represents the intent-to-treat (ITT) population. The number analyzed per row represents participants with data at each time point.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Part 1 - Inclisiran | Part 1 - Placebo
Number analyzed (Participants) | 19 | 37
Percentage Change
  Day 90: number analyzed (Participants) | 18 | 37
  Day 90 | 41.2 (243.94) | 42.0 (170.41)
  Day 150: number analyzed (Participants) | 17 | 34
  Day 150 | 230.8 (640.11) | 126.9 (380.15)
  Day 180: number analyzed (Participants) | 18 | 31
  Day 180 | 115.1 (490.17) | 45.2 (143.24)

46. Secondary Outcome: Percent Change in High-Sensitivity C-Reactive Protein (hsCRP) From Baseline to Subsequent Visits up to Day 720: Part 2
Description: Percentage change in hsCRP from baseline to subsequent visits up to Day 720
Time Frame: Baseline, Days 330, 510 ,690, 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
Percentage Change
  Day 330: number analyzed (Participants) | 15 | 25
  Day 330 | 178.9 (657.67) | 17.3 (73.29)
  Day 510: number analyzed (Participants) | 16 | 30
  Day 510 | 266.7 (936.76) | 64.7 (204.54)
  Day 690: number analyzed (Participants) | 13 | 22
  Day 690 | 29.0 (125.18) | 37.5 (92.40)
  Day 720: number analyzed (Participants) | 17 | 27
  Day 720 | 49.6 (167.16) | 38.60 (112.57)

47. Secondary Outcome: Absolute Change in High-Sensitivity C-Reactive Protein (hsCRP) From Baseline to Subsequent Visits up to Day 180: Part 1
Description: Absolute Change in High-Sensitivity C-Reactive Protein (hsCRP) from Baseline to subsequent visits up to Day 180
Time Frame: Baseline, Days 90, 150, 180
Population: as for outcome 45
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
mg/L
  Day 90: number analyzed (Participants) | 18 | 37
  Day 90 | -3.2 (9.46) | 0.7 (4.25)
  Day 150: number analyzed (Participants) | 17 | 34
  Day 150 | 0.5 (15.07) | 1.1 (6.51)
  Day 180: number analyzed (Participants) | 18 | 31
  Day 180 | -3.8 (9.33) | 0.2 (3.75)

48. Secondary Outcome: Absolute Change in High-Sensitivity C-Reactive Protein (hsCRP) From Baseline to Subsequent Visits up to Day 720: Part 2
Description: Absolute Change in High-Sensitivity C-Reactive Protein (hsCRP) from baseline to subsequent visits up to Day 720
Time Frame: Baseline, Days 330, 510, 690, 720
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Part 2 - Placebo-Inclisiran | Part 2 - Inclisiran-Inclisiran
Number analyzed (Participants) | 19 | 34
mg/L
  Day 330: number analyzed (Participants) | 15 | 25
  Day 330 | -4.0 (9.98) | -0.4 (2.81)
  Day 510: number analyzed (Participants) | 16 | 30
  Day 510 | -3.4 (10.07) | 0.9 (4.75)
  Day 690: number analyzed (Participants) | 13 | 22
  Day 690 | -4.7 (10.21) | 0.7 (3.94)
  Day 720: number analyzed (Participants) | 17 | 27
  Day 720 | -3.7 (9.86) | -0.2 (4.25)

49. Secondary Outcome: Percent Change in Apo-B From Baseline to Day 150
Description: Percentage change in Apo-B from baseline to Day 150 as demonstrated using the ANCOVA statisitical model.
Time Frame: Baseline, Day 150
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Percentage change | 3.55 [-13.60 to 20.71] | -0.75 [-11.50 to 9.99]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Test type: Superiority; p = 0.6814, ANCOVA; Mean Difference (Final Values) = -4.31, 95% CI 2-sided [-24.88 to 16.27]

50. Secondary Outcome: Percent Change in Non-HDL-C From Baseline to Day 150
Description: Percentage Change in non-HDL-C from baseline to Day 150 as demonstrated using the ANCOVA statisitical model.
Time Frame: Baseline, Day 150
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Percentage Change | 2.46 [-19.12 to 24.05] | 0.37 [-12.68 to 13.42]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Test type: Superiority; p = 0.8725, ANCOVA; Mean Difference (Final Values) = -2.10, 95% CI 2-sided [-27.70 to 23.51]

51. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Day 150
Description: Percentage change in total cholesterol from baseline to Day 150 as demonstrated using the ANCOVA statisitical model.
Time Frame: Baseline, Day 150
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 19 | 37
Percentage Change | 1.51 [-16.49 to 19.50] | 0.71 [-10.39 to 11.82]
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Test type: Superiority; p = 0.9425, ANCOVA; Mean Difference (Final Values) = -0.79, 95% CI 2-sided [-22.30 to 20.72]

52. Secondary Outcome: Proportion of Subjects With ≥30% LDL-C Reduction of From Baseline at Day 150
Description: Number of participants in each group with ≥30% LDL-C reduction from baseline at Day 150 using the Regression Logistic Statistical Model
Time Frame: Baseline, Day 150
Population: ITT Population: All participants randomized into the study comprised the intent-to-treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 - Placebo | Part 1 - Inclisiran
Number analyzed (Participants) | 18 | 34
Participants | 3 | 6
Statistical Analysis 1: Comparison: Part 1 - Placebo vs Part 1 - Inclisiran; Test type: Superiority; Regression, Logistic; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.2 to 5.2]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of approximately 2 years.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Groups:
- Part 1: Inclisiran: Participants who received a dose of 300 milligram (mg) Inclisiran for injection administered by SC injection on Day 1 and Day 90.
- Part 1: Placebo: Participants who received a dose of placebos administered by SC injection on Day 1 and Day 90.
- Part 1:All Patients: Total of all patients
- Part 2: Inclisiran: Participants who received a dose of 300 mg inclisiran for injection administered by SC injection on Day 270, Day 450 and Day 630.
Arm/Group | Part 1: Inclisiran | Part 1: Placebo | Part 1:All Patients | Part 2: Inclisiran
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/19 | 0/56 | 3/53
Serious Adverse Events (participants affected / at risk) | 2/37 | 1/19 | 3/56 | 11/53
Other Adverse Events (participants affected / at risk) | 12/37 | 6/19 | 18/56 | 29/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Inclisiran (N=37) | Part 1: Placebo (N=19) | Part 1:All Patients (N=56) | Part 2: Inclisiran (N=53)
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 2
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 1 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Family stress (Social circumstances) | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Inclisiran (N=37) | Part 1: Placebo (N=19) | Part 1:All Patients (N=56) | Part 2: Inclisiran (N=53)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 2
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 0 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 1
Goitre (Endocrine disorders) | 0 | 0 | 0 | 1
Scleral haemorrhage (Eye disorders) | 1 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Gastrooesophageal sphincter insufficiency (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 2 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Allergy to arthropod bite (Immune system disorders) | 1 | 0 | 1 | 0
Bacterial vulvovaginitis (Infections and infestations) | 0 | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 4
Genitourinary chlamydia infection (Infections and infestations) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 2
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection viral (Infections and infestations) | 2 | 2 | 4 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 1 | 2 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Ureaplasma infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 2
Alanine aminotransferase abnormal (Investigations) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1 | 1
Blood 25-hydroxycholecalciferol decreased (Investigations) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 2
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 3
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 1 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Cardiac valve prosthesis user (Social circumstances) | 0 | 0 | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT03851705/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT03851705/SAP_001.pdf